CLINICAL TRIAL: NCT04553705
Title: Impact of Different Treatment Modalities on Immunity Against COVID-19
Brief Title: Omega-3, Nigella Sativa, Indian Costus, Quinine, Anise Seed, Deglycyrrhizinated Licorice, Artemisinin, Febrifugine on Immunity of Patients With (COVID-19)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Collaborators: Maternity and Children Hospital, Makkah (Other); University of Arizona (Other)
Responsible Party: Principal Investigator, Mohamed Medhat Abdelwahab Gamaleldin, Clinical researcher, Beni-Suef University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TQ/Omega-3 on COVID-19; DOI: 10.31219/osf.io/u56fc (Other: OSFPREPRINTS- MAY-4/2020)
Record Dates: First submitted 2020-09-15; First posted 2020-09-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Covid19; Immunodeficiency
Keywords: COVID-19; omega3; thymoquinone
MeSH Terms: conditions — COVID-19; Immunologic Deficiency Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Omega-3/thymoquinone supplementation (Experimental): 10 patients that will receive every 14-days Omega-3/thymoquinone supplementation (300-400mg EPA & 200-300mg DHA) (3% thymoquinone) per day for one month.
  In addition to the standard care
  Interventions: Drug: Omega 3/Nigella Sativa Oil
- Omega-3/thymoquinone / Indian Costus supplementation (Experimental): 10 patients that will receive every 14-days Omega-3/thymoquinone supplementation (300-400mg EPA & 200-300mg DHA), (3% thymoquinone),(Indian Costus) per day for one month.
  In addition to the standard care
  Interventions: Drug: Omega 3/Nigella Sativa Oil/Indian Costus
- Omega-3/thymoquinone / Quinine pills (Experimental): 10 patients that will receive every 14-days Omega-3/thymoquinone supplementation (300-400mg EPA & 200-300mg DHA), (3% thymoquinone),(1g Quinine) per day for one month.
  In addition to the standard care
  Interventions: Drug: Omega 3/Nigella Sativa Oil/Quinine pills
- Omega-3/thymoquinone / Anise seed capsule (Experimental): 10 patients that will receive every 14-days Omega-3/thymoquinone supplementation (300-400mg EPA & 200-300mg DHA), (3% thymoquinone),(450mg anise seed) per day for one month.
  In addition to the standard care
  Interventions: Drug: Omega 3/Nigella Sativa Oil/Anise seed capsule
- Omega-3/thymoquinone / Deglycyrrhizinated Licorice (Experimental): 10 patients that will receive every 14-days Omega-3/thymoquinone supplementation (300-400mg EPA & 200-300mg DHA), (3% thymoquinone),(Deglycyrrhizinated Licorice 800 mg ) per day for one month.
  In addition to the standard care
  Interventions: Drug: Omega 3/Nigella Sativa Oil/Deglycyrrhizinated Licorice
- Active Comparator: standard care (Active Comparator): The standard protocol care for COVID-19 approved from ministry of health at Saudi arabia
  Interventions: Drug: Active Comparator

INTERVENTIONS:
Drug: Omega 3/Nigella Sativa Oil — Omega-3 supplementation 1000mg contains (300-400mg EPA & 200-300mg DHA)
  Nigella sativa supplementation (1g black seed oil contain 3% thymoquinone
  Arms: Omega-3/thymoquinone supplementation
Drug: Omega 3/Nigella Sativa Oil/Indian Costus — Omega-3 supplementation 1000mg contains (300-400mg EPA & 200-300mg DHA)
  Nigella sativa supplementation (1g black seed oil contain 3% thymoquinone
  Indian Costus supplements
  Arms: Omega-3/thymoquinone / Indian Costus supplementation
Drug: Omega 3/Nigella Sativa Oil/Quinine pills — Omega-3 supplementation 1000mg contains (300-400mg EPA & 200-300mg DHA)
  Nigella sativa supplementation (1g black seed oil contain 3% thymoquinone
  Quinine supplementation (1g Quinine)
  Arms: Omega-3/thymoquinone / Quinine pills
Drug: Omega 3/Nigella Sativa Oil/Anise seed capsule — Omega-3 supplementation 1000mg contains (300-400mg EPA & 200-300mg DHA)
  Nigella sativa supplementation (1g black seed oil contain 3% thymoquinone
  Anise seed supplementation (450mg anise seed)
  Arms: Omega-3/thymoquinone / Anise seed capsule
Drug: Omega 3/Nigella Sativa Oil/Deglycyrrhizinated Licorice — Omega-3 supplementation 1000mg contains (300-400mg EPA & 200-300mg DHA)
  Nigella sativa supplementation (1g black seed oil contain 3% thymoquinone
  Deglycyrrhizinated Licorice 800 mg
  Arms: Omega-3/thymoquinone / Deglycyrrhizinated Licorice
Drug: Active Comparator — Standard protocol care of COVID-19 infection
  Arms: Active Comparator: standard care

SUMMARY:
The first version of this preprint article is registered on the 4th of May 2020 under the digital object identifier of:10.31219/osf.io/u56fc.

COVID-19 infections virus spread worldwide and impact many countries with sever economical sequences. The effective antiviral medication or vaccination for the virus is unavailable until the present date and it takes months or years to discover the effective treatment or test the efficacy of the discovered treatment.

Based on these facts, the human immune system against the virus may have an effective role to regulate the infection and reduce the mortality rate among the infected patients. This proposed research article aims to explore the available medication/ natural supplementation to boost the immunity system of the patients against COVID-19 infections and reduce the mortality rate among infected patients. Methods: a proposed clinical trial will be carried out to investigate the effect of the different treatment modalities on the human immune system against COVID-19 infection.

DETAILED DESCRIPTION:
Natural supplementations have many reported effects on the human health ranged from immunity boosting to effective antiviral effect. Omeg-3 as an example affect the human health by many mechanisms e.g. Anti-oxidant, immunity boosting agent. Moreover, Omega-3 exerts an antiviral effect on Flu virus by inhibiting influenza virus replication 1. On the other hand, black seed supplementation exerts a chelation effect on sickle cell anemia patients and inhibits Human Heme Metabolism 2. Moreover, black seed exerts an antiviral effect on the replication of old coronavirus and the expression of (TRP-genes) family 3. In addition, Omega-3 regulates the human immunity against bacterial and viral infections 4. During the past years, many natural sources exerts an antimalarial effect with perfect reported results 5.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic with respiratory or systemic symptoms
* Positive nasopharyngeal swab for COVID-19
* CT imaging showing viral pneumonia
* Temperature 38°C
* Respiratory rate < 25 /min
* Oxygen saturation (pulse oximetry) >95%

Exclusion Criteria:

* Pregnant or breast feeding
* Hepatic failure Child-Pugh C
* Negative swab test of (SARS)-(CoV-2)
* Expected life is less than 24 hours
* End-stage lung disease

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2021-12-04 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | 30 Days
  Time to Clinical recovery
Recovery rate from positive to negative swaps | 14 Days
  Percentage of patients returned to negative swaps of COVID-19
Fever to normal temperature in days | 15 Days
  Number of days for fever remission T=37.5°C
Remission of lung inflammation in CT or X-ray | 30 Days
  Number of days to report lungs recovery in chest X ray or CT
Length of hospitalization | 10 Days
  Number of days for hospitalization
(PCR levels) polymerase chain reaction assay levels | 10 Days
  Change of (PCR levels) > 50% in comparison with PCR levels at the admission
Respiratory indexes | 10 Days
  P O2/Fi O2 which reflects patients' oxygen saturation
C-reactive protein mg/L | 25 Days
  C-reactive protein milligrams per deciliter correlated with inflammation
Serum Ferritin ng/ml | 25 Days
  Serum Ferritin Nanograms per milliliter correlated with iron overload and illness severity
Lactic acid dehydrogenase U/L | 25 Days
  Lactic acid dehydrogenase unit per litter correlated with illness severity
leukocytes count μl | 30 Days
  leukocytes in microliter correlated with mortality
Lipid profile [LDL, HDL, Total cholesterol ] | 14 Days
  Mg/dl correlated with lipid peroxidation that linked to oxidative stress
total plasma antioxidant capacity | 14 Days
  Evaluate the antioxidant response against the free radicals produced in COVID-19 infection measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: HASSAN Masmali [consultant of Pediatrics], M.D, Study Director — Maternity and Children hospital,Mecca, Saudi Arabia; MOHAMED M ABDELWAHAB GAMALELDIN, Ph.D Candidate, Principal Investigator — Beni-Suef University, Faculty of Pharmacy; SHAIMAA M Nashat SAYED ABDELHALIM, Ph.D Candidate, Principal Investigator — Beni-Suef University, Faculty of Pharmacy
Locations (1):
- Maternity and Children hospital, Mecca, Mecca Region, Saudi Arabia